CLINICAL TRIAL: NCT05172310
Title: PET Imaging of Tumors in Pancreas, Bile Ducts, Stomach and Ovaries by a Novel Tracer, 68Ga-FAPI-46 = Fibroblast Activation Protein Inhibitor
Brief Title: PET Imaging of Solid Tumors by a Novel Tracer, 68Ga-FAPI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rimma Axelsson, Professor, Karolinska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H035-FAPI; 2020-002568-30 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Epithelial Ovarian Cancer
Keywords: 68-Ga FAPI; PET/CT; Pancreatic Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Fibroblast activating protein inhibitor; FAPI; Epithelial Ovarian Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Carcinoma, Ovarian Epithelial | interventions — FAPI-46; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Investigators select subjects that are scheduled for
  * surgical removal of either a malignant lesion in the pancreas, bile ducts, or stomach (first arm)
  * surgical removal of primary stage epithelial cancer of the ovary (EOC), interval debulking surgery (IDS) of EOC or surgical removal/tissue biopsy of recurrent EOC (first arm)
  * surgical removal of a benign lesion in the pancreas (second arm)
  All patients will undergo a PET/CT with the interventional drug/radiotracer 68Ga-FAPI-46 before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients (Experimental): * Adults with suspected cancer of either pancreas, bile ducts or stomach
  * Adults with primary and recurrent epithelial ovarian cancer (EOC)
  Interventions: Drug: 68Ga-FAPI-46; Device: PET/CT
- Non cancer patients (Active Comparator): Non cancer patients operated for non-malignant diseases in pancreas during the same period of time will be investigated with the same procedure.
  Interventions: Drug: 68Ga-FAPI-46; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-FAPI-46 — * [68Ga] Ga-FAPI-46 Solution for Injection is manufactured at the Karolinska University Hospital Radiopharmacy facilities, for imaging studies with Positron Emission Tomography (PET).
  * It is a radiolabelled Fibroblast Activation Protein Inhibitor (FAPI) used for PET of a number of different cancer entities.
  * Depending on the labelling yield 50 - 370 megabecquerel (MBq) of [68Ga] Ga-FAPI-46 Solution for Injection will be administered intravenously 60 minutes prior to whole-body PET image acquisition.
Device: PET/CT — * Combined PET and computed tomography (CT) imaging with 68Ga-FAPI-46 will be performed using the same protocol on a "Biograph 6" PET/CT scanner (Siemens, Erlangen, Germany) and "General Electrics" (GE) Discovery 710, Milwaukee, Wisconsin, USA at the Department of Nuclear Medicine, Karolinska Huddinge within 2 weeks before surgery.
  * PET/CT imaging will be performed in dynamic mode at one bed position centered over the primary tumor for 45 minutes.
  * At 60 minutes post injection, a whole-body PET will be acquired.

SUMMARY:
Cancers of the pancreas, bile ducts, stomach and ovaries are dismal diseases with most patients being diagnosed in advanced stages leading to a bad prognosis. These cancers can be difficult to diagnose and sometimes impossible to differentiate from underlying benign conditions. Establishing the correct diagnosis of primary cancer lesions and possible spread to other organs in time is pivotal for choosing the right therapy. Routinely applied staging procedures are however not always reliable. The main aim in this study is to evaluate the diagnostic accuracy of PET/CT with a novel radiotracer, FAPI, in the primary diagnosis of cancers in the pancreas, stomach and bile ducts as well as in patients with primary and recurrent epithelial ovarian cancer (EOC).

DETAILED DESCRIPTION:
Malignant tumors exceeding 1-2 mm in size require formation of a supporting stroma, which includes vascular cells, inflammatory cells and fibroblasts . Several organs in the upper gastro-intestinal tract are known to develop tumors with strong desmoplastic reaction characterized by pervasive growth of tumor stroma. The pancreas, stomach, bile ducts and ovaries are all organs with this property. Within tumor stroma, a subpopulation of fibroblasts called cancer-associated fibroblasts (CAFs) are known to be involved in growth, migration and progression of the tumor.

The Fibroblast Activation Protein (FAP) is one of the more prominent stroma markers and was the focus in the development of an agent for imaging and, eventually, even targeted radionuclide therapy. FAP is a type II membrane bound glycoprotein absent or only expressed at insignificant levels, in normal tissues in adults. The FAP inhibitor, FAPI, gets selectively enriched in tissues where its target protein is expressed and there is no or very limited FAPI uptake in all normal organs. This opens new possibilities for the detection of malignant lesions with higher stromal content based on the high contrast positron emission tomography (PET) images obtained with a 68-Gallium (68Ga) radiolabeled - FAPI compound. As cancers in pancreas, stomach, bile ducts and ovaries are all characterized by abundant desmoplasia that constitutes up to 90% of the total tumor volume and contains extracellular matrix, immune cells, vasculature and CAFs, it would be suitable for targeted imaging with FAPI.

Preliminary studies show elevated FAPI uptake in many tumors rich in fibroblasts along with low background uptake. The main objective of this prospective study is to improve non-invasive diagnostics of malignancy in tumors of pancreas, stomach, bile ducts and ovaries, all known for a strong desmoplastic reaction by evaluating the diagnostic accuracy of PET/CT with a novel radiotracer, FAPI in the primary diagnosis and staging of such cancers.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for surgical removal of either a pancreatic, biliary or gastric lesion.

  - Consecutive patients scheduled for primary surgical removal of early stage epithelial ovarian cancer (EOC), interval debulking surgery of EOC or surgical removal or tissue biopsy of recurrent EOC
* Signed informed consent.

Common Exclusion Criteria for all study populations:

* Age ≤18 year
* Pregnancy and lactation
* Significantly reduced renal function
* Allergy to iodinated contrast media
* Subjects that for some reason are unable to exercise their own rights, such as cognitive function impairment.

Additional Exclusion Criteria for study populations with either pancreatic-, gastric or bile duct cancer:

• Known metastatic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of FAPI-PET/CT in primary tumors | up to 18 months
  To validate the proportion of false-positive and false-negative FAPI-PET/CT findings in primary pancreas, biliary and gastric tumors as well as in primary and recurrent EOC with postsurgical or true cut biopsy histopathological confirmation of diagnosis (PAD) as a reference standard

SECONDARY OUTCOMES:
Diagnostic accuracy of FAPI-PET/CT in metastases | up to 18 months
  To validate the proportion of false-positive and false-negative FAPI-PET/CT findings in resected metastatic tumor tissue/resected lymph nodes, in primary (and recurrent for EOC) tumors, by using postsurgical tissue samples or biopsies as well as PAD as a reference standard.
Immunohistochemistry | up to 18 months
  To investigate the correlation between in-vivo uptake of FAPI and ex-vivo immunohistochemically determined biomarker expression in the stroma of these tumors (both benign and malignant) with PAD as a reference standard
FAPI-PET/CT and stroma markers as prognostic factors for Disease Free Survival (DFS) | up to 5 years
  Disease Free Survival (DFS) at 1-year, 2-years and 5-years clinical follow-ups.
FAPI-PET/CT and stroma markers as prognostic factors for Overall Survival (OS) | up to 5 years
  Overall Survival (OS) at 1-year, 2-years and 5-years clinical follow-ups.
Correlation between FAPI-PET/CT imaging results and those of conventional radiology | up to 18 months
  To investigate the difference in diagnostic accuracy of FAPI-PET/CT compared to conventional imaging diagnostics performed according to clinical routine, by using postsurgical PAD as a reference standard both for differentiation between malignant and benign lesions as well as for N and M staging.
Safety of 68Ga-FAPI-46 | up to 1 month
  Frequency of
  * Adverse Events (AEs)
  * Adverse Reactions (ARs)-
  * Serious Adverse Events (SAEs) and
  * Suspected Unexpected Serious Adverse Reactions (SUSARs).

CONTACTS AND LOCATIONS:
Overall Officials: Rimma Axelsson, Professor, Principal Investigator — Medical Radiation Physics and Nuclear Medicine, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson B, Goldberg I, Kopolovic J. Inflammatory response in cervical intraepithelial neoplasia and squamous cell carcinoma of the uterine cervix. Pathol Res Pract. 1997;193(7):491-5. doi: 10.1016/s0344-0338(97)80102-1. PMID 9342755
- [Background] Whatcott CJ, Posner RG, Von Hoff DD, Han H. Desmoplasia and chemoresistance in pancreatic cancer. In: Grippo PJ, Munshi HG, editors. Pancreatic Cancer and Tumor Microenvironment. Trivandrum (India): Transworld Research Network; 2012. Chapter 8. Available from http://www.ncbi.nlm.nih.gov/books/NBK98939/ PMID 22876390
- [Background] Moon SB, Hur JM, Koo HH, Suh YL, Shin HB, Seo JM, Lee SK. Desmoplastic small round cell tumor of the stomach mimicking a gastric cancer in a child. J Korean Surg Soc. 2011 Jun;80 Suppl 1(Suppl 1):S80-4. doi: 10.4174/jkss.2011.80.Suppl1.S80. Epub 2011 Jun 17. PMID 22066092
- [Background] Baba AI, Câtoi C. TUMORS OF THE ALIMENTARY SYSTEM [Internet]. The Publishing House of the Romanian Academy; 2007 [cited 2020 Apr 1]. Available from: https://www.ncbi.nlm.nih.gov/books/NBK9565/
- [Background] Fiori ME, Di Franco S, Villanova L, Bianca P, Stassi G, De Maria R. Cancer-associated fibroblasts as abettors of tumor progression at the crossroads of EMT and therapy resistance. Mol Cancer. 2019 Mar 30;18(1):70. doi: 10.1186/s12943-019-0994-2. PMID 30927908
- [Background] Ham IH, Lee D, Hur H. Role of Cancer-Associated Fibroblast in Gastric Cancer Progression and Resistance to Treatments. J Oncol. 2019 Jun 9;2019:6270784. doi: 10.1155/2019/6270784. eCollection 2019. PMID 31281359
- [Background] Ma Y, Zhu J, Chen S, Li T, Ma J, Guo S, Hu J, Yue T, Zhang J, Wang P, Wang X, Chen G, Liu Y. Activated gastric cancer-associated fibroblasts contribute to the malignant phenotype and 5-FU resistance via paracrine action in gastric cancer. Cancer Cell Int. 2018 Jul 20;18:104. doi: 10.1186/s12935-018-0599-7. eCollection 2018. PMID 30038550
- [Background] Ohlund D, Handly-Santana A, Biffi G, Elyada E, Almeida AS, Ponz-Sarvise M, Corbo V, Oni TE, Hearn SA, Lee EJ, Chio II, Hwang CI, Tiriac H, Baker LA, Engle DD, Feig C, Kultti A, Egeblad M, Fearon DT, Crawford JM, Clevers H, Park Y, Tuveson DA. Distinct populations of inflammatory fibroblasts and myofibroblasts in pancreatic cancer. J Exp Med. 2017 Mar 6;214(3):579-596. doi: 10.1084/jem.20162024. Epub 2017 Feb 23. PMID 28232471
- [Background] Brivio S, Cadamuro M, Strazzabosco M, Fabris L. Tumor reactive stroma in cholangiocarcinoma: The fuel behind cancer aggressiveness. World J Hepatol. 2017 Mar 28;9(9):455-468. doi: 10.4254/wjh.v9.i9.455. PMID 28396716
- [Background] Olive KP, Jacobetz MA, Davidson CJ, Gopinathan A, McIntyre D, Honess D, Madhu B, Goldgraben MA, Caldwell ME, Allard D, Frese KK, Denicola G, Feig C, Combs C, Winter SP, Ireland-Zecchini H, Reichelt S, Howat WJ, Chang A, Dhara M, Wang L, Ruckert F, Grutzmann R, Pilarsky C, Izeradjene K, Hingorani SR, Huang P, Davies SE, Plunkett W, Egorin M, Hruban RH, Whitebread N, McGovern K, Adams J, Iacobuzio-Donahue C, Griffiths J, Tuveson DA. Inhibition of Hedgehog signaling enhances delivery of chemotherapy in a mouse model of pancreatic cancer. Science. 2009 Jun 12;324(5933):1457-61. doi: 10.1126/science.1171362. Epub 2009 May 21. PMID 19460966
- [Background] Hingorani SR, Harris WP, Beck JT, Berdov BA, Wagner SA, Pshevlotsky EM, Tjulandin SA, Gladkov OA, Holcombe RF, Korn R, Raghunand N, Dychter S, Jiang P, Shepard HM, Devoe CE. Phase Ib Study of PEGylated Recombinant Human Hyaluronidase and Gemcitabine in Patients with Advanced Pancreatic Cancer. Clin Cancer Res. 2016 Jun 15;22(12):2848-54. doi: 10.1158/1078-0432.CCR-15-2010. Epub 2016 Jan 26. PMID 26813359
- [Background] Park JE, Lenter MC, Zimmermann RN, Garin-Chesa P, Old LJ, Rettig WJ. Fibroblast activation protein, a dual specificity serine protease expressed in reactive human tumor stromal fibroblasts. J Biol Chem. 1999 Dec 17;274(51):36505-12. doi: 10.1074/jbc.274.51.36505. PMID 10593948
- [Background] Scanlan MJ, Raj BK, Calvo B, Garin-Chesa P, Sanz-Moncasi MP, Healey JH, Old LJ, Rettig WJ. Molecular cloning of fibroblast activation protein alpha, a member of the serine protease family selectively expressed in stromal fibroblasts of epithelial cancers. Proc Natl Acad Sci U S A. 1994 Jun 7;91(12):5657-61. doi: 10.1073/pnas.91.12.5657. PMID 7911242
- [Background] Egger C, Cannet C, Gerard C, Suply T, Ksiazek I, Jarman E, Beckmann N. Effects of the fibroblast activation protein inhibitor, PT100, in a murine model of pulmonary fibrosis. Eur J Pharmacol. 2017 Aug 15;809:64-72. doi: 10.1016/j.ejphar.2017.05.022. Epub 2017 May 12. PMID 28506908
- [Background] Tillmanns J, Hoffmann D, Habbaba Y, Schmitto JD, Sedding D, Fraccarollo D, Galuppo P, Bauersachs J. Fibroblast activation protein alpha expression identifies activated fibroblasts after myocardial infarction. J Mol Cell Cardiol. 2015 Oct;87:194-203. doi: 10.1016/j.yjmcc.2015.08.016. Epub 2015 Aug 28. PMID 26319660
- [Background] Moir JA, Mann J, White SA. The role of pancreatic stellate cells in pancreatic cancer. Surg Oncol. 2015 Sep;24(3):232-8. doi: 10.1016/j.suronc.2015.05.002. Epub 2015 May 19. PMID 26080604
- [Background] Laverman P, van der Geest T, Terry SY, Gerrits D, Walgreen B, Helsen MM, Nayak TK, Freimoser-Grundschober A, Waldhauer I, Hosse RJ, Moessner E, Umana P, Klein C, Oyen WJ, Koenders MI, Boerman OC. Immuno-PET and Immuno-SPECT of Rheumatoid Arthritis with Radiolabeled Anti-Fibroblast Activation Protein Antibody Correlates with Severity of Arthritis. J Nucl Med. 2015 May;56(5):778-83. doi: 10.2967/jnumed.114.152959. Epub 2015 Apr 9. PMID 25858044
- [Background] van der Geest T, Laverman P, Gerrits D, Walgreen B, Helsen MM, Klein C, Nayak TK, Storm G, Metselaar JM, Koenders MI, Boerman OC. Liposomal Treatment of Experimental Arthritis Can Be Monitored Noninvasively with a Radiolabeled Anti-Fibroblast Activation Protein Antibody. J Nucl Med. 2017 Jan;58(1):151-155. doi: 10.2967/jnumed.116.177931. Epub 2016 Aug 4. PMID 27493266
- [Background] Meletta R, Muller Herde A, Chiotellis A, Isa M, Rancic Z, Borel N, Ametamey SM, Kramer SD, Schibli R. Evaluation of the radiolabeled boronic acid-based FAP inhibitor MIP-1232 for atherosclerotic plaque imaging. Molecules. 2015 Jan 27;20(2):2081-99. doi: 10.3390/molecules20022081. PMID 25633335
- [Background] Watabe T, Liu Y, Kaneda-Nakashima K, Shirakami Y, Lindner T, Ooe K, Toyoshima A, Nagata K, Shimosegawa E, Haberkorn U, Kratochwil C, Shinohara A, Giesel F, Hatazawa J. Theranostics Targeting Fibroblast Activation Protein in the Tumor Stroma: 64Cu- and 225Ac-Labeled FAPI-04 in Pancreatic Cancer Xenograft Mouse Models. J Nucl Med. 2020 Apr;61(4):563-569. doi: 10.2967/jnumed.119.233122. Epub 2019 Oct 4. PMID 31586001
- [Background] Jansen K, Heirbaut L, Cheng JD, Joossens J, Ryabtsova O, Cos P, Maes L, Lambeir AM, De Meester I, Augustyns K, Van der Veken P. Selective Inhibitors of Fibroblast Activation Protein (FAP) with a (4-Quinolinoyl)-glycyl-2-cyanopyrrolidine Scaffold. ACS Med Chem Lett. 2013 Mar 18;4(5):491-6. doi: 10.1021/ml300410d. eCollection 2013 May 9. PMID 24900696
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Meyer C, Dahlbom M, Lindner T, Vauclin S, Mona C, Slavik R, Czernin J, Haberkorn U, Calais J. Radiation Dosimetry and Biodistribution of 68Ga-FAPI-46 PET Imaging in Cancer Patients. J Nucl Med. 2020 Aug;61(8):1171-1177. doi: 10.2967/jnumed.119.236786. Epub 2019 Dec 13. PMID 31836685
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Löhr JM, Kordes M, Rutkowski W, Heuchel R, Gustafsson-Liljefors M, Russom A, et al. Overcoming diagnostic issues in precision treatment of pancreatic cancer. Expert Rev Precis Med Drug Dev. 2018 May 4;3(3):189-95.
- [Background] Micke P, Ostman A. Exploring the tumour environment: cancer-associated fibroblasts as targets in cancer therapy. Expert Opin Ther Targets. 2005 Dec;9(6):1217-33. doi: 10.1517/14728222.9.6.1217. PMID 16300472
- [Background] Neesse A, Bauer CA, Ohlund D, Lauth M, Buchholz M, Michl P, Tuveson DA, Gress TM. Stromal biology and therapy in pancreatic cancer: ready for clinical translation? Gut. 2019 Jan;68(1):159-171. doi: 10.1136/gutjnl-2018-316451. Epub 2018 Sep 3. PMID 30177543
- [Background] Guggenheim DE, Shah MA. Gastric cancer epidemiology and risk factors. J Surg Oncol. 2013 Mar;107(3):230-6. doi: 10.1002/jso.23262. Epub 2012 Nov 5. PMID 23129495
- [Background] Yashiro M, Hirakawa K. Cancer-stromal interactions in scirrhous gastric carcinoma. Cancer Microenviron. 2010 Jan 26;3(1):127-35. doi: 10.1007/s12307-010-0036-5. PMID 21209779
- [Background] Kirstein MM, Vogel A. Epidemiology and Risk Factors of Cholangiocarcinoma. Visc Med. 2016 Dec;32(6):395-400. doi: 10.1159/000453013. Epub 2016 Dec 1. PMID 28229073
- [Background] Zhang H, Zhu J, Ke F, Weng M, Wu X, Li M, Quan Z, Liu Y, Zhang Y, Gong W. Radiological Imaging for Assessing the Respectability of Hilar Cholangiocarcinoma: A Systematic Review and Meta-Analysis. Biomed Res Int. 2015;2015:497942. doi: 10.1155/2015/497942. Epub 2015 Sep 1. PMID 26448940
- [Background] Anderson CD, Rice MH, Pinson CW, Chapman WC, Chari RS, Delbeke D. Fluorodeoxyglucose PET imaging in the evaluation of gallbladder carcinoma and cholangiocarcinoma. J Gastrointest Surg. 2004 Jan;8(1):90-7. doi: 10.1016/j.gassur.2003.10.003. PMID 14746840
- [Background] Olthof SC, Othman A, Clasen S, Schraml C, Nikolaou K, Bongers M. Imaging of Cholangiocarcinoma. Visc Med. 2016 Dec;32(6):402-410. doi: 10.1159/000453009. Epub 2016 Dec 6. PMID 28229074
- [Background] Vaquero J, Aoudjehane L, Fouassier L. Cancer-associated fibroblasts in cholangiocarcinoma. Curr Opin Gastroenterol. 2020 Mar;36(2):63-69. doi: 10.1097/MOG.0000000000000609. PMID 31934895
- [Background] Itou RA, Uyama N, Hirota S, Kawada N, Wu S, Miyashita S, Nakamura I, Suzumura K, Sueoka H, Okada T, Hatano E, Tsutsui H, Fujimoto J. Immunohistochemical characterization of cancer-associated fibroblasts at the primary sites and in the metastatic lymph nodes of human intrahepatic cholangiocarcinoma. Hum Pathol. 2019 Jan;83:77-89. doi: 10.1016/j.humpath.2018.08.016. Epub 2018 Aug 30. PMID 30172911
- [Background] Loktev A, Lindner T, Burger EM, Altmann A, Giesel F, Kratochwil C, Debus J, Marme F, Jager D, Mier W, Haberkorn U. Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention. J Nucl Med. 2019 Oct;60(10):1421-1429. doi: 10.2967/jnumed.118.224469. Epub 2019 Mar 8. PMID 30850501
- [Background] Giesel FL, Kratochwil C, Lindner T, Marschalek MM, Loktev A, Lehnert W, Debus J, Jager D, Flechsig P, Altmann A, Mier W, Haberkorn U. 68Ga-FAPI PET/CT: Biodistribution and Preliminary Dosimetry Estimate of 2 DOTA-Containing FAP-Targeting Agents in Patients with Various Cancers. J Nucl Med. 2019 Mar;60(3):386-392. doi: 10.2967/jnumed.118.215913. Epub 2018 Aug 2. PMID 30072500
- [Background] Sharma P, Singh SS, Gayana S. Fibroblast Activation Protein Inhibitor PET/CT: A Promising Molecular Imaging Tool. Clin Nucl Med. 2021 Mar 1;46(3):e141-e150. doi: 10.1097/RLU.0000000000003489. PMID 33351507
- [Background] Zhang L, Sanagapalli S, Stoita A. Challenges in diagnosis of pancreatic cancer. World J Gastroenterol. 2018 May 21;24(19):2047-2060. doi: 10.3748/wjg.v24.i19.2047. PMID 29785074
- [Background] Shrikhande SV, Barreto SG, Goel M, Arya S. Multimodality imaging of pancreatic ductal adenocarcinoma: a review of the literature. HPB (Oxford). 2012 Oct;14(10):658-68. doi: 10.1111/j.1477-2574.2012.00508.x. Epub 2012 Jun 14. PMID 22954001